CLINICAL TRIAL: NCT01798719
Title: Low Glycemic Index Mediterranean Diet Effect on Moderate or Severe Non-alcoholic Fatty Liver Disease
Brief Title: Effect of Mediterranean Diet on Non-alcoholic Fatty Liver Disease
Acronym: Nutriepa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Alberto R Osella, Senior Researcher, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPINUT3
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: NAFLD
Keywords: NAFLD; Clinical Trial; Mediterranean Diet; Low Glycemic Index
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet: Dietary Advice (Placebo Comparator): Some general dietary advice about healthy dietary components, servings size and frequency of servings
  Interventions: Behavioral: General Advice
- Low glycemic index Mediterranean Diet (Experimental): Low glycemic index Mediterranean Diet prescription with indication about type of foods than can be consumed frequently (green foods), sometimes (yellow foods) and never (red foods)
  Interventions: Behavioral: Low Glycemic Index Mediterranean Diet

INTERVENTIONS:
Behavioral: Low Glycemic Index Mediterranean Diet — A list of foods that may be consumed frequently (green foods), sometimes (yellow foods) and never (red foods)
  Arms: Low glycemic index Mediterranean Diet
Behavioral: General Advice — Only general advice about diet
  Arms: Diet: Dietary Advice

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a clinical/biochemical condition associated with the metabolic syndrome. As the disease stems from excess calorie intake and lack of physical activity, the correction of unhealthy lifestyles is the background of any prevention and treatment strategy

DETAILED DESCRIPTION:
The majority of NAFLD patients are characterized by high body mass index, insulin resistance and they show a remarkably higher energy intake in comparison to individuals without hepatic steatosis. Several authors have proposed dietary weight loss strategies to ameliorate or reverse fatty liver because of the potential role of weight loss on the supposed risk factors of liver injury, mainly insulin resistance, free fatty acid levels, and pro-inflammatory and profibrotic adipokines. There are no definite data regarding how much and how rapidly weight loss should be to have the more favorable effects, but in obese children, the larger the weight loss, the larger the decrease of liver enzyme levels and the lower the prevalence of NAFLD. The American Gastroenterological Association recommends a weight loss target of 10% of baseline. A loss of at least 10% of body weight in obese patients is associated with a normalization of previously abnormal liver function tests as well as decreased hepatomegaly, but even a moderate weight loss (approximately 6% of baseline weight) can improve insulin resistance and intrahepatic liver content.

ELIGIBILITY:
Inclusion Criteria:

* Subject enrolled in the cohort Nutriep assembled in 2005-2007
* Moderate or severe NAFLD

Exclusion Criteria:

* Middle NAFLD
* Not enrolled in the Nutriep cohort
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Non-alcoholic Fatty Liver Disease Ultrasonography Score | Six months
  A semiquantitative score to measure Non-alcoholic Fatty Liver Disease will be used

CONTACTS AND LOCATIONS:
Overall Officials: Alberto R Osella, MD, PhD, Principal Investigator — IRCCS Saverio de Bellis; Giovanni Misciagna, MD, PhD, Study Director — IRCCS Saverio de Bellis
Locations (1):
- Laboratory of Epidemiology and Biostatistics, IRCCS Saverio de Bellis, Castellana Grotte, BA, Italy

REFERENCES:
- [Background] Cozzolongo R, Osella AR, Elba S, Petruzzi J, Buongiorno G, Giannuzzi V, Leone G, Bonfiglio C, Lanzilotta E, Manghisi OG, Leandro G; NUTRIHEP Collaborating Group; Donnaloia R, Fanelli V, Mirizzi F, Parziale L, Crupi G, Detomaso P, Labbate A, Zizzari S, Depalma M, Polignano A, Lopinto D, Daprile G. Epidemiology of HCV infection in the general population: a survey in a southern Italian town. Am J Gastroenterol. 2009 Nov;104(11):2740-6. doi: 10.1038/ajg.2009.428. Epub 2009 Jul 28. PMID 19638964
- [Derived] Hooper L, Abdelhamid AS, Jimoh OF, Bunn D, Skeaff CM. Effects of total fat intake on body fatness in adults. Cochrane Database Syst Rev. 2020 Jun 1;6(6):CD013636. doi: 10.1002/14651858.CD013636. PMID 32476140
- [Derived] Misciagna G, Del Pilar Diaz M, Caramia DV, Bonfiglio C, Franco I, Noviello MR, Chiloiro M, Abbrescia DI, Mirizzi A, Tanzi M, Caruso MG, Correale M, Reddavide R, Inguaggiato R, Cisternino AM, Osella AR. Effect of a Low Glycemic Index Mediterranean Diet on Non-Alcoholic Fatty Liver Disease. A Randomized Controlled Clinici Trial. J Nutr Health Aging. 2017;21(4):404-412. doi: 10.1007/s12603-016-0809-8. PMID 28346567